CLINICAL TRIAL: NCT04088136
Title: Enhancing Older Adults' Everyday Memory Function
Brief Title: Everyday Memory Intervention
Acronym: EMMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H19341; 1R21AG059942-01A1 (NIH)
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Aging
Keywords: everyday memory; ecological momentary assessment; memory complaint; metacognition; mnemonics; external aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Everyday Metacognitive Memory (Experimental): Training in techniques for managing memory demands in everyday life
  Interventions: Behavioral: Everyday Metacognitive Memory Intervention
- Memory Strategy Control (Active Comparator): Trains the use of memory strategies for learning new associations and concepts
  Interventions: Behavioral: Memory Strategy Control Intervention

INTERVENTIONS:
Behavioral: Everyday Metacognitive Memory Intervention — Provides training in use of techniques and procedures to enhance proactive self-regulatory control over everyday memory demands, including strategies for learning information, planning for meeting everyday goals, and monitoring of efficacy of goal pursuit.
  Arms: Everyday Metacognitive Memory
Behavioral: Memory Strategy Control Intervention — Trains use of standard mnemonic techniques such as imagery and sentence generation for learning new associations and organizational and distinctiveness-based strategies for learning sets of items (e.g., word lists).
  Arms: Memory Strategy Control

SUMMARY:
Evaluates an intervention designed to improve everyday memory function, contrasting people receiving the intervention with a group that receives traditional memory strategy training.

DETAILED DESCRIPTION:
This project seeks to develop and validate a novel approach to training everyday memory functioning in older adults. The approach (1) trains people to use simple but effective memory skills that have broad applicability in everyday life and (2) shapes a set of skills and habits of mind that will increase the likelihood of effective use of skills and memory aids. It is based on a metacognitive perspective on self-regulation in cognitively demanding situations and informed by recent theories about how suboptimal habit patterns can be altered. The approach has not yet been used in an everyday memory intervention in high-functioning, community-dwelling older adults. The proposed research validates ecological momentary assessment methods to get actual behavioral measures of forgetting in everyday life. It then uses these procedures in a randomized experiment that contrasts the everyday memory intervention group with a traditional memory-strategy training group. The hypothesis is that the everyday memory training intervention will reduce everyday memory errors and memory complaints, whereas the memory strategy training will alter strategy use and memory performance, with little cross-over effect. The hypothesized pattern will establish the explicit benefits of our everyday memory intervention procedures and demonstrate the limitation of standard memory training for that purpose.

ELIGIBILITY:
Inclusion Criteria:

* 70 - 85 years of age
* in fair to good health
* free of major neurocognitive impairment
* English speaking
* endorsed Smartphone and computer users (or willing to learn)

Exclusion Criteria:

* diagnosis of any major neurological problems (e.g. stroke, Parkinson's disease, dementia)
* 1.5 SD below age-normed mean (or lower) on the TICS
* low computer and smart phone literacy
* and poor self-rated health.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hertzog, Ph.D, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Adult Cognition Lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey H, Dunlosky J, Hertzog C. Metacognitive training at home: does it improve older adults' learning? Gerontology. 2010;56(4):414-20. doi: 10.1159/000266030. Epub 2009 Dec 11. PMID 20016124
- [Background] Bailey HR, Dunlosky J, Hertzog C. Does strategy training reduce age-related deficits in working memory? Gerontology. 2014;60(4):346-56. doi: 10.1159/000356699. Epub 2014 Feb 27. PMID 24577079
- [Background] Bottiroli S, Cavallini E, Dunlosky J, Vecchi T, Hertzog C. The importance of training strategy adaptation: a learner-oriented approach for improving older adults' memory and transfer. J Exp Psychol Appl. 2013 Sep;19(3):205-18. doi: 10.1037/a0034078. Epub 2013 Aug 26. PMID 23978160
- [Background] Bottiroli S, Cavallini E, Dunlosky J, Vecchi T, Hertzog C. Self-guided strategy-adaption training for older adults: Transfer effects to everyday tasks. Arch Gerontol Geriatr. 2017 Sep;72:91-98. doi: 10.1016/j.archger.2017.05.015. Epub 2017 Jun 7. PMID 28609674
- [Background] Dunlosky J, Cavallini E, Roth H, McGuire CL, Vecchi T, Hertzog C. Do self-monitoring interventions improve older adult learning? J Gerontol B Psychol Sci Soc Sci. 2007 Jun;62 Spec No 1:70-6. doi: 10.1093/geronb/62.special_issue_1.70. PMID 17565167
- [Background] Dunlosky J, Hertzog C. Measuring strategy production during associative learning: the relative utility of concurrent versus retrospective reports. Mem Cognit. 2001 Mar;29(2):247-53. doi: 10.3758/bf03194918. PMID 11352207
- [Background] Dunlosky, J., Hertzog, C., Kennedy, M. R. T., & Thiede, K. W. (2005). The self-monitoring approach for effective learning. Cognitive Technology, 10, 4-11.
- [Background] Dunlosky J, Kubat-Silman AK, Hertzog C. Training monitoring skills improves older adults' self-paced associative learning. Psychol Aging. 2003 Jun;18(2):340-5. doi: 10.1037/0882-7974.18.2.340. PMID 12825781
- [Background] Hertzog C, McGuire CL, Horhota M, Jopp D. Does believing in "use it or lose it" relate to self-rated memory control, strategy use, and recall? Int J Aging Hum Dev. 2010;70(1):61-87. doi: 10.2190/AG.70.1.c. PMID 20377166
- [Background] Hertzog C, Sinclair SM, Dunlosky J. Age differences in the monitoring of learning: cross-sectional evidence of spared resolution across the adult life span. Dev Psychol. 2010 Jul;46(4):939-48. doi: 10.1037/a0019812. PMID 20604613
- [Background] Hertzog C, Dunlosky J. Metacognition in Later Adulthood: Spared Monitoring Can Benefit Older Adults' Self-regulation. Curr Dir Psychol Sci. 2011 Jun;20(3):167-173. doi: 10.1177/0963721411409026. PMID 24478539
- [Background] Hertzog C, Lineweaver TT, Hines JC. Computerized assessment of age differences in memory beliefs. Percept Mot Skills. 2014 Oct;119(2):609-28. doi: 10.2466/03.10.PMS.119c23z4. Epub 2014 Sep 26. PMID 25259780
- [Background] Hertzog C, Lustig E, Pearman A, Waris A. Behaviors and Strategies Supporting Everyday Memory in Older Adults. Gerontology. 2019;65(4):419-429. doi: 10.1159/000495910. Epub 2019 Feb 8. PMID 30739118
- [Background] Lineweaver, T. T., & Hertzog, C. (1998). Adults' efficacy and control beliefs regarding memory and aging: Separating general from personal beliefs. Aging, Neuropsychology, and Cognition 5, 264-296. doi: 10.1076/anec.5.4.264.771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was converted to a completely on-line study due to the COVID-19 pandemic. Enrollment began in March of 2021.
Period: Overall Study
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Started | 35 | 33
Completed | 30 | 32
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Adults ages 70-85 from greater Atlanta GA area meeting inclusion/exclusion criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 non-response
  years
    number analyzed (Participants) | 35 | 32 | 67
    (all) | 76.3 (4.8) | 75.2 (4.6) | 75.8 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 nonresponse
  Participants
    number analyzed (Participants) | 34 | 33 | 67
    Female | 21 | 19 | 40
    Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 31 | 33 | 64
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — questionnaire self-report
  Participants
    American Indian or Alaska Native | 1 | 1 | 2
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
    Black or African American | 4 | 5 | 9
    White | 26 | 26 | 52
    More than one race | 2 | 0 | 2
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 33 | 68
AB5C Personality Scales [Mean (Standard Deviation); unit: units on a scale] — Big 5 personality facets. Scaled as average item Likert endorsement (1-7 scale). Higher scores indicate greater self-rated attribute (e.g., higher conscientiousness). Population: one participant did not complete the AB5C inventory
  units on a scale
    AB5C Gregariousness: number analyzed (Participants) | 34 | 33 | 67
    AB5C Gregariousness | 3.2 (0.7) | 2.9 (0.6) | 3.1 (0.7)
    AB5C Stability: number analyzed (Participants) | 34 | 33 | 67
    AB5C Stability | 3.5 (0.6) | 3.4 (0.7) | 3.5 (0.6)
    AB5C Understanding: number analyzed (Participants) | 34 | 33 | 67
    AB5C Understanding | 4.4 (0.4) | 4.4 (0.5) | 4.4 (0.4)
    AB5C Introspection: number analyzed (Participants) | 34 | 33 | 67
    AB5C Introspection | 3.7 (0.7) | 4.0 (0.5) | 3.9 (0.6)
    AB5C Conscientiousness: number analyzed (Participants) | 34 | 33 | 67
    AB5C Conscientiousness | 3.9 (0.5) | 4.1 (0.4) | 4.0 (0.5)
Victoria Activity Scale [Mean (Standard Deviation); unit: units on a scale] — Augmented Victoria Activity Scale (total) Scaled as average Likert item response (1-7 scale; higher scores indicate more activity) Population: one nonresponse
  units on a scale
    number analyzed (Participants) | 34 | 33 | 67
    (all) | 4.2 (0.6) | 4.1 (0.6) | 4.1 (0.6)
Pattern Comparison Test [Mean (Standard Deviation); unit: scores on a scale] — Pattern Comparison Test is a measure of processing speed. Respondents are asked to quickly determine whether two stimuli are the same or different. A sum score reflecting the total number of correct responses is calculated for each respondent. The minimum score is 0 and the maximum possible score is 60. Higher scores reflect more correct responses. More correct responses indicate faster processing speed. Population: missing data due to program failure during remote administration
  scores on a scale
    number analyzed (Participants) | 34 | 30 | 64
    (all) | 16.1 (4.3) | 14.8 (5.6) | 15.5 (4.9)
Shipley Vocabulary Test [Mean (Standard Deviation); unit: scores on a scale] — Shipley Vocabulary Test is a measure of vocabulary and is used as a measure of crystallized ability. Respondents are shown a word and asked to identify a synonym out of a list of options. A sum score reflecting the total number of correct responses is calculated for each respondent. The minimum score is 0 and the maximum possible score is 40. Higher scores reflect more correct responses. More correct responses indicate better crystallized ability. Population: missing data due to program failure during remote administration
  scores on a scale
    number analyzed (Participants) | 34 | 32 | 66
    (all) | 34.3 (3.4) | 35.7 (3.1) | 35.0 (3.3)
ETS Letter Sets Test [Mean (Standard Deviation); unit: scores on a scale] — Educational Testing Services (ETS) Letter Sets Test is a measure of fluid intelligence. Each item has five sets of letters with four letters in each set. Four of the sets are alike in some way while one set is not alike. Respondents are asked to indicate which set does not belong in each item. A sum score reflecting the total number of correct responses is calculated for each respondent. The minimum score is 0 and the maximum possible score is 30. Higher scores reflect more correct responses. More correct responses indicate better fluid ability. Population: missing data due to program failure during remote administration
  scores on a scale
    number analyzed (Participants) | 34 | 32 | 66
    (all) | 8.9 (2.5) | 9.1 (3.3) | 9.0 (2.9)
Mobile Device Proficiency Questionnaire (MDPQ-16) [Mean (Standard Deviation); unit: units on a scale] — Self-report questionnaire focused on an individual's ability to perform different tasks with a mobile device. Sub-scales include: mobile device basics, communication, data and file storage, internet, calendar, entertainment, privacy, and troubleshooting and software management. The mean was calculated for each subscale and then summed to compute the total score. Higher scores indicate individuals can more easily use different functions of a mobile device. Sub-scale ranges 1 = Never tried, 5 = Very easily. The total score ranges from a minimum of 8 to a maximum of 40. Population: missing questionnaires
  units on a scale
    number analyzed (Participants) | 33 | 33 | 66
    (all) | 31.5 (7.2) | 31.8 (6.4) | 31.7 (6.8)
Technology Experience Profile [Mean (Standard Deviation); unit: units on a scale] — Self-report questionnaire assessed the frequency with which people use different types of technology. The individual scales include: communication technology, computer technology, everyday technology, health technology, recreational technology, and transportation technology. The mean was calculated for each subscale and then were summed to compute the total score. Higher scores indicate individuals use different types of technology more frequently. Sub-scale ranges from 1 = Not sure what it is, 5 = Used frequently. The total score ranges from a minimum of 6 to a maximum of 30. Population: missing questionnaire
  units on a scale
    number analyzed (Participants) | 34 | 33 | 67
    (all) | 23.1 (2.1) | 23.4 (2.4) | 23.2 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Everyday Memory Failures
Description: Across the data collection period, participants audio recorded descriptions of their memory failures on a smartphone app. The audio recordings were transcribed and then cleaned and qualitatively coded so that the number of memory failures each participant reported during the data collection period could be counted. The data was qualitatively coded to ensure an accurate count of the number of memory failures per participant without counting duplicate events or accidental reports. Average daily number of reported memory failures from EMA & daily diaries is reported.
Time Frame: minimum 8 day period after training on app prior to posttest
Measure: Mean (Standard Error); unit: average daily number memory failures/day
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 30 | 32
average daily number memory failures/day | 0.55 (0.57) | 0.62 (0.71)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; Test type: Equivalence — A one-tailed independent samples t-test was conducted. A p-value of .05 was used to determine statistical significance; p = .67, t-test, 2 sided; Use of pooled error term, df = 60; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.42 to 0.55], Standard Error of Mean 0.17 — Negative number reflects fewer errors in EMMI group, as predicted

2. Primary Outcome: Prospective Memory Lab Contacts
Description: Number of successfully completed lab contacts (maximum of 4)
Time Frame: Two weeks prior to posttest
Measure: Mean (Standard Error); unit: number of contacts
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 30 | 32
number of contacts | 2.8 (0.2) | 3.0 (0.2)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; Test type: Superiority — Everyday Metacognitive Memory group predicted to have superior scores to Memory Strategy Control; p < .47, t-test, 1 sided; Mean Difference (Final Values) = -0.20, Standard Error of Mean 0.28 — pooled error term, equal variance assumption, df = 60

3. Primary Outcome: Prospective Memory Lab Contact Efficiency
Description: median absolute time deviation (in minutes) from scheduled lab contact for completed contacts
Time Frame: Two weeks prior to posttest
Population: data only available for persons who successfully completed at least one laboratory contact
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 29 | 31
minutes | 4.4 (1.7) | 4.2 (1.1)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; Test type: Superiority; p < .13, t-test, 1 sided; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-3.7 to 7.6], Standard Error of Mean 2.0

4. Primary Outcome: Everyday Cognition Simulation Task: ATM Task (Number of Errors)
Description: Computerized task to simulate use of an ATM machine. Measure: number of errors
Time Frame: posttest only
Measure: Mean (Standard Error); unit: number of errors
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 25 | 28
number of errors | 9.08 (0.79) | 10.14 (1.59)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; Test type: Equivalence — Directional hypothesis of fewer errors in Everyday Metacognitive Memory group; p = .57, t-test, 2 sided — A p-value of .05 was used to determine statistical significance; Pooled error term, df = 51; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-4.8 to 2.6], Standard Error of Mean 1.8

5. Primary Outcome: Czaja Everyday Cognition Simulation Task: Prescription Refill Task (Number of Errors)
Description: Computerized task to simulate use of an automated telephone program to refill prescriptions. Measure: Number of errors
Time Frame: posttest only
Population: Missing data caused by program run-time errors aborting program without recording results for several participants (6 Everyday Metacognitive Memory; 5 Memory Strategy Control)
Measure: Mean (Standard Error); unit: number of errors
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 24 | 27
number of errors | 9.29 (1.74) | 8.44 (1.55)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; Test type: Equivalence — Two-tailed test of hypothesis of fewer errors in EMMI group; p = .72, t-test, 2 sided — A p-value of .05 was used to determine statistical significance; Pooled error term, df = 49; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-3.8 to 5.5], Standard Error of Mean 2.3

6. Primary Outcome: Free Recall Test
Description: Computerized task to present 30 concrete nouns, 6 from 5 taxonomic categories (Hultsch, Hertzog, Dixon, & Small, 1998) Measure is proportion of 30 words recalled
Time Frame: pretest and posttest (approximately 1 month lag)
Population: One missing case due to program failure when administering the test
Measure: Mean (Standard Error); unit: proportion of words recalled
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 29 | 32
proportion of words recalled
  Pretest | 0.27 (0.05) | 0.31 (0.05)
  Posttest | 0.37 (0.05) | 0.44 (0.05)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; We ran a 2 X 2 (Group X Time) mixed model analysis with repeated measures on Time (pretest, posttest). Hypothesis was that Memory Strategy Control group would show greater improvements from pretest to posttest in recall scores; Test type: Other — Test of Group X Time interaction; p < .69, Mixed Models Analysis; pooled df = 59

7. Primary Outcome: Associative Recall Test
Description: Computerized task to present 40 concrete-concrete associatively unrelated noun pairs (Hertzog, Sinclair, & Dunlosky, 2010) Outcome is proportion of 40 words correctly recalled.
Time Frame: pretest and posttest (approximately 1 month lag)
Measure: Mean (Standard Error); unit: proportion of words recalled
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 30 | 32
proportion of words recalled
  Pretest | 0.52 (0.04) | 0.53 (0.04)
  Posttest | 0.55 (0.04) | 0.66 (0.04)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; We ran a 2 X 2 (Group X Time) mixed effect model with repeated measures on Time (pretest-posttest). Predicted hypothesis was greater pretest-posttest improvement in the Memory Strategy Contol group; Test type: Other — One-tailed test of Group X Time interaction; p < .037, Mixed Models Analysis

8. Primary Outcome: Story Recall
Description: gist recall of narrative story (total number of propositions (ideas) from story recalled)
Time Frame: posttest only
Measure: Mean (Standard Error); unit: number of ideas recalled
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 30 | 31
number of ideas recalled | 30.8 (1.6) | 29.7 (1.9)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; Test type: Other; p = .69, t-test, 2 sided; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-4.0 to 8.4], Standard Error of Mean 9.9 — one instance of missing data due to computer failure during testing. Pooled error term resulting in df = 59

9. Primary Outcome: Everyday Cognition Simulation Task: ATM Task (Time in Seconds)
Description: Computerized task to simulate use of an ATM machine. Measure: time to complete task (in seconds)
Time Frame: posttest only
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 25 | 28
seconds | 852.10 (61.74) | 902.10 (80.53)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; Test type: Equivalence — Directional hypothesis of shorter time in Everyday Metacognitive Memory group; p = .63, t-test, 2 sided — A p-value of .05 was used to determine statistical significance; Use of pooled error term, DF = 51; Mean Difference (Final Values) = -50.0, 95% CI 2-sided [-257.4 to 157.4], Standard Error of Mean 103.3

10. Primary Outcome: Czaja Everyday Cognition Simulation Task: Prescription Refill Task (Time in Seconds)
Description: Computerized task to simulate use of an automated telephone program to refill prescriptions. Measure: time to complete task (in seconds)
Time Frame: posttest only
Population: as for outcome 5
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 24 | 27
seconds | 590.50 (31.68) | 579.90 (30.15)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; Test type: Equivalence — Two-tailed test of hypothesis of shorter time in Everyday Metacognitive Memory group; p = .81, t-test, 2 sided — A p-value of .05 was used to determine statistical significance; Use of pooled error term, df = 49; Mean Difference (Final Values) = 10.6, 95% CI 2-sided [-77.4 to 98.5], Standard Error of Mean 43.8

11. Secondary Outcome: MFQ Memory Complaint (Frequency of Forgetting Scale)
Description: Summative Likert scale measuring frequency of reported memory problems for specific types of problems Measure is average item Likert rating on a 1-7 scale. Higher score indicates fewer memory problems
Time Frame: pretest and posttest (approximately 1 month lag)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 30 | 32
units on a scale
  Pretest | 4.9 (0.2) | 5.1 (0.2)
  Posttest | 5.0 (0.2) | 5.0 (0.2)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; We conducted a 2 X 2 (Group X Time) mixed effects model with repeated measures on Time (pretest, posttest). Hypothesis was greater reduction in memory complaints from pretest to posttest in EMMI group; Test type: Other; p < .14, Mixed Models Analysis; mixed procedure with unrestricted error covariance matrix. Pooled df for MSWithin = 60

12. Secondary Outcome: PBMI Specific Memory Self-Efficacy
Description: The Personal Beliefs about Memory Instruments (PBMI) Specific Memory Self-Efficacy measurement is a summative visual analog rating scale measuring self-rated memory aggregated over multiple specific types of memory. Outcomes scaled in average proportion of distance from left (0) to maximum of 1.00 (higher scores indicate greater memory self-efficacy).
Time Frame: pretest and posttest (approximately 1 month lag)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 30 | 32
units on a scale
  Pretest | 0.65 (0.02) | 0.71 (0.02)
  Posttest | 0.72 (0.02) | 0.73 (0.02)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; We ran a 2 X 2 (Group X Time) mixed effect model with repeated measures on Time (pretest-posttest); Test type: Other; p = .037, Mixed Models Analysis

13. Secondary Outcome: PBMI Memory Control
Description: Summative visual analog rating scale measuring self-rated control over everyday. Outcome is scaled as average proportion of maximum endorsement (ranging from 0 to 1.0, with higher scores indicate greater perceived control)
Time Frame: pretest and posttest (approximately 1 month lag)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 30 | 32
units on a scale
  Pretest | 0.79 (0.03) | 0.80 (0.03)
  Posttest | 0.90 (0.02) | 0.89 (0.02)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; We ran a 2 X 2 (Group X Time) mixed effects model with repeated measures on Time (pretest, posttest); Test type: Other — Hypothesis was greater increase in memory self-efficacy for Everyday Metacognitive Memory group; p < .33, Mixed Models Analysis; mixed model specified unrestricted residual (error) covariance matrix. Pooled df in MS Error = 60

14. Secondary Outcome: MCQ Internal Scale
Description: Summative Likert scale obtaining self-rated frequency of use of internal mnemonic strategies in everyday life. Average Likert rating on 1-5 scale (higher scores indicate greater use of strategies)
Time Frame: pretest and posttest (approximately 1 month lag)
Measure: Mean (Standard Error); unit: average units on a scale
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 30 | 32
average units on a scale
  Pretest | 1.92 (0.12) | 2.01 (0.11)
  Posttest | 2.31 (0.11) | 2.26 (0.11)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; We ran a 2 X 2 (Group X Time) mixed effects model with repeated measures on Time (pretest, posttest). Hypothesis was greater increase in memory control in EMMI group; Test type: Other; p < .20, Mixed Models Analysis

15. Secondary Outcome: MCQ External
Description: Summative Likert scale obtaining self-rated frequency of use of external memory aids. Outcome is scaled as average Likert rating on 1-5 scale. Higher score indicates greater use of external aids.
Time Frame: pretest and posttest (approximately 1 month lag)
Measure: Mean (Standard Error); unit: average units on a scale
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
Number analyzed (Participants) | 30 | 32
average units on a scale
  Pretest | 3.34 (0.09) | 3.28 (0.09)
  Posttest | 3.38 (0.08) | 3.30 (0.08)
Statistical Analysis 1: Comparison: Everyday Metacognitive Memory vs Memory Strategy Control; Test type: Other — Hypothesis was greater increase in use of external mnemonics in EMMI group; p < .20, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Everyday Metacognitive Memory | Memory Strategy Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32

LIMITATIONS AND CAVEATS:
We were forced to change the protocol to allow only remote participation from home given the COVID-19 pandemic. Adjusting assessment procedures took time and also forced us to reduce the scope of the intervention, especially one on one shaping of trained procedures, given constraints on available staff to coach participants with an accelerated testing schedule. Changes in assessment procedures led to some lost data through failed programs or participant errors in saving data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT04088136/Prot_001.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT04088136/SAP_002.pdf
  • Informed Consent Form (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT04088136/ICF_000.pdf